CLINICAL TRIAL: NCT00217425
Title: Bevacizumab and CHOP (A-CHOP) in Combination for Patients With Peripheral T-Cell or Natural Killer Cell Neoplasms
Brief Title: Bevacizumab and Combination Chemotherapy in Treating Patients With Peripheral T-Cell Lymphoma or Natural Killer Cell Neoplasms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000441194; U10CA021115 (NIH); E2404 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma
Keywords: anaplastic large cell lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; peripheral T-cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Peripheral | interventions — Bevacizumab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (A-CHOP followed by MA) (Experimental): Patients receive 6-8 cycles of bevacizumab and combination chemotherapy comprising cyclophosphamide, doxorubicin, vincristine, and prednisone (A-CHOP) followed by 8 cycles of maintenance bevacizumab (MA), as outlined below. Bevacizumab 15 mg/kg is administered on day 1 over 90 min (first cycle), 60 min (second cycle) and 30 min for the subsequent cycles. CHOP (cyclophosphamide 750 mg/m 2 ; doxorubicin 50 mg/m 2 ; vincristine 1.4 mg/m2 [max. 2 mg]; prednisone 100 mg daily on days 1-5) is administered on day 1 of a 21-day cycle. Radiographic response is assessed after cycles 3, 6 and 8 of ACHOP and after cycle 8 of MA. Patients receive six cycles of ACHOP if they achieve a complete response (CR) after three cycles, eight cycles if they achieve a partial response (PR) after three cycles. Non-responders are removed from the study. ACHOP responders receive maintenance bevacizumab 15 mg/kg every 21 days for eight cycles.
  Interventions: Biological: bevacizumab; Drug: cyclophosphamide; Drug: doxorubicin; Drug: prednisone; Drug: vincristine

INTERVENTIONS:
Biological: bevacizumab — A - CHOP: 15 mg/kg IV infusion once every 21 days for 6-8 cycles. Bevacizumab is to be administered prior to CHOP therapy. Continuous bevacizumab: 15 mg/kg IV infusion once every 21 days.
  Initial dose should be infused over 90 minutes. If no adverse reactions occur, the second dose should be administered over 60 minutes. Again, if no adverse reactions occur, the third and subsequent doses should be administered over 30 minutes. If infusion-related adverse reactions occur, subsequent infusions should be administered over the shortest period that is well-tolerated. Infusions should be run in via a volumetric infusion device. Do NOT administer as an IV push or bolus.
  Other Names: NSC 704865,; RhuMAb VEGF,; Recombinant Humanized Monoclonal Anti-VEGF Antibody.
Drug: cyclophosphamide — IV infusion per institutional guidelines.
  Other Names: Cytoxan,; Neosar,; CTX,; CPM.
Drug: doxorubicin — Intravenously, either as a bolus injection or as a continuous infusion through a central venous line.
  Other Names: Adriamycin, Rubex, Adriamycin RDF, Adriamycin PFS, hydroxydaunorubicin,; hydroxydaunomycin, ADR.
Drug: prednisone — Prednisone is taken orally.
  Other Names: Deltasone,; Orasone,; Medicorten,; Panasol-S,; Liquid-Pred.
Drug: vincristine — IV push using extravasation precautions.
  Other Names: Oncovin,; Vincasar PFS vincristine sulfate,; VCR,; leucocristine,; LCR.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Bevacizumab may also stop the growth of cancer cells by blocking blood flow to the cancer. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with several chemotherapy drugs (combination chemotherapy) works in treating patients with peripheral T-cell lymphoma or natural killer cell neoplasms.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 12-month progression-free survival of patients with peripheral T-cell or natural killer cell neoplasms treated with bevacizumab and combination chemotherapy comprising cyclophosphamide, doxorubicin, vincristine, and prednisone (A-CHOP).

Secondary

* Determine the overall response rate (complete remission [CR, unconfirmed CR, or functional CR] and partial remission) in these patients after courses 3, 6, and 8 of this treatment regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive 6-8 cycles of A-CHOP followed by 8 cycles of maintenance bevacizumab (MA), as outlined below. Bevacizumab 15 mg/kg is administered on day 1 over 90 min (first cycle), 60 min (second cycle) and 30 min for the subsequent cycles. CHOP (cyclophosphamide 750 mg/m 2 ; doxorubicin 50 mg/m 2 ; vincristine 1.4 mg/m2 [max. 2 mg]; prednisone 100 mg daily on days 1-5) is administered on day 1 of a 21-day cycle. Radiographic response is assessed after cycles 3, 6 and 8 of ACHOP and after cycle 8 of MA. Patients receive six cycles of ACHOP if they achieve a complete response (CR) after three cycles, eight cycles if they achieve a partial response (PR) after three cycles. Non-responders are removed from the study. ACHOP responders receive maintenance bevacizumab 15 mg/kg every 21 days for eight cycles.

After completion of study treatment, patients are followed every 3 months for 2 years, and then every 6 months for up to 5 years.

PROJECTED ACCRUAL: A total of 43 patients will be accrued for this study within 22 months.

ACTUAL ACCRUAL: 46

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnosis of peripheral T-cell or natural killer cell neoplasm

  * Any stage disease allowed
  * HTLV-positive tumors allowed
* At least one objective measurable disease parameter. Abnormal positron emission tomography scans are not considered evidence of measurable disease unless results are confirmed by CT scan or other appropriate imaging techniques
* Age 18 and over
* ECOG Performance status 0-2
* Absolute neutrophil count ≥ 1,000/mm^3(500/mm^3 if due to bone marrow involvement with lymphoma)
* Platelet count ≥ 100,000/mm^3(50,000/mm^3 if due to bone marrow involvement with lymphoma)
* Bilirubin ≤ 2.0 mg/dL (≤ 3 times upper limit of normal [ULN] if due to hepatic involvement with lymphoma)
* AST ≤ 2 times ULN (5 times ULN if due to hepatic involvement with lymphoma)
* PT, INR, and PTT ≤ 1.5 times normal
* Creatinine ≤ 2.0 mg/dL
* Urinary protein:creatinine ratio ≤ 1
* History of deep venous thrombosis allowed provided patient is on a stable dose of anticoagulants for at least 2 weeks prior to study entry
* LVEF ≥ 50%
* History of pulmonary embolism allowed provided patient is on a stable dose of anticoagulants for at least 2 weeks prior to study entry
* One prior cycle of CHOP for PTCL allowed
* More than 4 weeks since prior major invasive surgery or open biopsy
* At least 7 days since prior minor surgery. Peripheral lymph node core biopsy, bone marrow biopsy, fine needle aspiration, skin biopsy, or central line placement are not considered minor surgical procedures
* More than 7 days since prior and no concurrent anti-platelet drugs (e.g., ticlopidine, clopidogrel, or cilostazol) except aspirin or other nonsteroidal anti-inflammatory drugs
* Concurrent anticoagulants allowed provided patient is on a stable dose

  * INR must be stable for at least 2 weeks prior to study entry
  * PT/INR and/or PTT must be closely monitored and levels kept within acceptable range for underlying thrombotic disease
  * Concurrent heparin flush for maintenance of central line patency allowed

EXCLUSION CRITERIA:

* Anaplastic lymphoma kinase (ALK)-positive T-cell large cell lymphoma. ALK-negative T-cell large cell lymphoma allowed
* Cutaneous T-cell lymphoma
* History of or current radiographic evidence of CNS metastasis, including previously treated, resected, or asymptomatic brain lesions or leptomeningeal involvement
* Evidence of bleeding diathesis or coagulopathy
* Cerebrovascular accident within the past 6 months
* Myocardial infarction within the past 6 months
* Unstable angina within the past 6 months
* New York Heart Association class II-IV congestive heart failure
* Uncontrolled hypertension (i.e., systolic blood pressure [BP] > 150 mm Hg or diastolic BP > 100 mm Hg)
* Other clinically significant cardiovascular or peripheral vascular disease
* Abdominal fistula within the past 6 months
* Gastrointestinal perforation within the past 6 months
* Intra-abdominal abscess within the past 6 months
* Concurrent major surgery
* Pregnant or nursing. Female patients must have negative pregnancy test. Fertile patients must use effective contraception
* History of active seizures
* Significant traumatic injury within the past 4 weeks
* Non-healing ulcer (unless involved with lymphoma)
* Bone fracture
* Active infection requiring parenteral antibiotics
* HIV positivity
* Other active malignancy within the past 6 months except carcinoma in situ of the cervix or basal cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-09-14 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen N. Ganjoo, MD, Study Chair — Veterans Affairs Medical Center - Palo Alto
Locations (110):
- United States (110):
  - California Cancer Care, Incorporated - Greenbrae, Greenbrae, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - La Grange Oncology Associates - Geneva, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Doylestown Hospital Cancer Center, Doylestown, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Central Pennsylvania Hematology and Medical Oncology Associates, PC, Lemoyne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was accrued on September 14, 2006.
Period: Overall Study
Arm/Group | Treatment (A-CHOP Followed by MA)
Started | 46
Treated | 44
Eligible and Treated | 39
Completed | 9
Not Completed | 37
Not completed — Never started treatment | 2
Not completed — Patient ineligible | 5
Not completed — Lack of Efficacy | 13
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 4
Not completed — Other complicating disease | 1
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Population: Eligible and treated
Arm/Group | Treatment (A-CHOP Followed by MA)
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 60 [21 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: 12-Month Progression-Free Survival (PFS)
Description: 12-month progression-free survival is defined as the probability of patients remaining alive and progression-free at 12 months from study entry.
Time Frame: Assessed every 3 months the first 2 years from study entry and every 6 months 3-5 years from study entry.
Population: Eligible and treated patients
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Treatment (A-CHOP Followed by MA)
Number analyzed (Participants) | 39
probability | 0.44 [.31 to .63]

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as proportion of patients who achieve complete remission [CR, unconfirmed CR (CRu) or Functional CR] or partial remission. Response is assessed using the criteria from the International Workshop to Standardize Criteria for Non-Hodgkin's Lymphoma (Chesen, 1999).
Time Frame: Assessed after cycle 3, cycle 6, and cycle 8 (if given).
Population: Eligible and treated
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Treatment (A-CHOP Followed by MA)
Number analyzed (Participants) | 39
proportion | 0.90 [0.76 to 0.93]

3. Secondary Outcome: 3-Year Overall Survival
Description: 3-year overall survival is defined as the probability of patients surviving at 3 years from study entry.
Time Frame: Assessed every 3 months the first 2 years from study entry and every 6 months 3-5 years from study entry.
Population: Eligible and treated patients
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Treatment (A-CHOP Followed by MA)
Number analyzed (Participants) | 39
probability | 0.39 [0.26 to 0.58]

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Groups:
- Treatment (ACHOP Followed by MA): Adverse events in all treated patients regardless of eligibility.
Arm/Group | Treatment (ACHOP Followed by MA)
Serious Adverse Events (participants affected / at risk) | 34/44
Other Adverse Events (participants affected / at risk) | 39/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (ACHOP Followed by MA) (N=44)
Anemia (Blood and lymphatic system disorders) | 3
White blood cell decreased (Investigations) | 14
Lymphocyte count decreased (Investigations) | 12
Neutrophil count decreased (Investigations) | 23
Platelet count decreased (Investigations) | 5
Ventricular arrhythmia (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 4
Restrictive cardiomyopathy (Cardiac disorders) | 1
Fatigue (General disorders) | 6
Weight loss (Investigations) | 1
Death NOS (General disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Colonic perforation (Gastrointestinal disorders) | 1
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Infections and infestations - Other, spe (Infections and infestations) | 2
Infections and infestations - Other, spe (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Anorectal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 4
Investigations - Other, specify (Investigations) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Vaginal inflammation (Reproductive system and breast disorders) | 1
Thromboembolic event (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (ACHOP Followed by MA) (N=44)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4
Anemia (Blood and lymphatic system disorders) | 15
White blood cell decreased (Investigations) | 7
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 7
Hypertension (Vascular disorders) | 5
Fatigue (General disorders) | 29
Fever (General disorders) | 4
Insomnia (Psychiatric disorders) | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Weight loss (Investigations) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 17
Nail loss (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 12
Constipation (Gastrointestinal disorders) | 14
Diarrhea (Gastrointestinal disorders) | 9
Abdominal distension (Gastrointestinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 9
Mucositis oral (Gastrointestinal disorders) | 13
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 15
Dysgeusia (Nervous system disorders) | 6
Vomiting (Gastrointestinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 6
Edema limbs (General disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Alkaline phosphatase increased (Investigations) | 6
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 19
Hypokalemia (Metabolism and nutrition disorders) | 6
Proteinuria (Renal and urinary disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 7
Investigations - Other, specify (Investigations) | 3
Dizziness (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 24
Watering eyes (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No